CLINICAL TRIAL: NCT05703516
Title: A Post Approval Commitment Study on Tabrecta® (Capmatinib) in South Korea; Open Label, Prospective, Multicenter, Post Approval Surveillance
Brief Title: A Post Approval Commitment Study on Tabrecta® (Capmatinib) in South Korea
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CINC280AKR01
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Non Small Cell Lung; Non Small Cell Lung Cancer; Non-small cell lung cancer; NSCLC; INC280; Non-small cell lung carcinoma (NSCLC); lung cancer; lung adenocarcinoma; Non small cell lung carcinoma; MET exon 14 deletion; METex14del; MET exon 14 skipping; MET exon 14 mutation; MET mutation; MET amplification; MET inhibitor; MET dysregulation; MET activation; MET signaling; MET pathway
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma of Lung | interventions — capmatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Capmatinib: Participants will be treated with capmatinib as per locally approved label
  Interventions: Other: Capmatinib

INTERVENTIONS:
Other: Capmatinib — There is no treatment allocation. Capmatinib will be prescribed by the physician as per locally approved label. Treatment duration depends on the decision of treating physician. No drug will be dispensed from Novartis
  Other Names: Tabrecta

SUMMARY:
This is an open label, prospective, multicenter, non-comparative study to assess the safety and effectiveness of Tabrecta® (Capmatinib) in real world setting. Also, this study is to fulfill the regulatory requirements as part of the RMP (Risk Management Plan) for Tabrecta® (Capmatinib), as requested by Korea Health Authority, MFDS (Ministry of Food and Drug Safety).

DETAILED DESCRIPTION:
The study is a post approval surveillance so there will be no comparator arm/drug nor blinding process.

Dose/regimen should follow locally approved label and it could be adjusted as per the decision from treating physician during treatment period, under their routine clinical practice. Treatment duration is deemed to the decision from treating physician under their routine clinical practice, since this study is a post approval surveillance and to look for safety profiles happening under real world practice. There will be no intervention from Novartis regarding dose/regimen and treatment duration.

This study will be completed after data collection of the last subject during the follow up period. The follow up period is recommended for up to 24 weeks after enrollment or up to the time of discontinuation of study drug (in case of early discontinuation) as per linical judgement of treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Subject who are diagnosed as exon 14 skipping mutated NSCLC from tissue or plasma(ctDNA) sample analysis by treating physician (i.e. Any kind of diagnostic methods the institution currently has. Diagnostic modalities for research purpose would be also allowable.)
* Subject who plan to receive Tabrecta® (Capmatinib) as per locally approved label

Exclusion Criteria:

* Subject with contraindication according to the locally approved label
* Subject whose medical record is not accessible
* Subject who are not willing to provide informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive Tabrecta® (Capmatinib) as per locally approved label.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs). | From date of first study dose to end of study, assessed up to approximately 28 weeks
  The number of participants with AEs and SAEs will be assessed

SECONDARY OUTCOMES:
Objective response rates (ORRs) assessed by investigator | Up to 24 weeks
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 and as assessed by the investigator.
Progression Free Survival (PFS) | Up to 24 weeks
  PFS defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- South Korea (9):
  - Novartis Investigative Site, Daegu, Dalseo Gu
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Daejeon
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Jeollanam
  - Novartis Investigative Site, Seoul

IPD SHARING:
Plan to Share IPD: No